CLINICAL TRIAL: NCT06444516
Title: A Single-Arm Study to Evaluate and Demonstrate Safety and Performance of a Novel Ocular Lubricant in Adult Subjects With Dry Eye Disease
Brief Title: Study of Safety and Performance of a Novel Ocular Lubricant in Subjects With Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEP918-C001
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FID123300 (Experimental): One drop of FID123300 ocular lubricant in each eye on Day 1 in the morning, followed by at least one drop in each eye 4 times a day on Days 2-30.
  Interventions: Other: FID123300 ocular lubricant

INTERVENTIONS:
Other: FID123300 ocular lubricant — Investigational ocular lubricant

SUMMARY:
The purpose of this study is to evaluate and demonstrate the efficacy and safety of an investigational ocular lubricant formulation in patients with mild to moderate dry eye disease (DED).

DETAILED DESCRIPTION:
The study will consist of a Screening visit, a Baseline visit on Day 1, a remote Compliance Check on Day 14, and an Exit visit on Day 30. The expected study duration of participation for each subject is 37 days, with 30 ± 5 days of exposure to the investigational product.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to understand and sign an approved informed consent form.
* Exhibit symptoms of dry eye at the Screening visit.
* Best Corrected Visual Acuity equal to or better than 20/80 Snellen in each eye at the Screening visit.
* Willing to discontinue use of all artificial tear supplements and use only the study product as directed starting at Visit 2/Day 1.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during the study.
* Ocular abnormalities that could adversely affect the safety or efficacy outcome.
* Uncontrolled active systemic diseases.
* Use of systemic medications known to cause dry eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Impact of Dry Eye on Everyday Life - Symptom Bother (IDEEL-SB) Questionnaire Score at Day 30 | Baseline (Day 1); Day 30
  The IDEEL-SB module consists of 20 questions that assess general dry eye symptoms a subject may experience. For each question, the subject will be instructed to select a single response that best represents their answer. The Symptom Bother score is calculated as the mean value of the non-missing item scores 1-20 multiplied by 25. A paired (one-sample) t-test will be used on the change from baseline value at Day 30 for hypothesis testing.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (9):
- United States (9):
  - Kindred Optics at Maitland Vision Center, Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Franklin Park Eye Center, PC, Franklin Park, Illinois
  - Kannarr Eye Care, LLC, Pittsburg, Kansas
  - SUNY College of Optometry Clinical Vision Research Center, New York, New York
  - ProCare Vision Center, Granville, Ohio
  - Wyomissing Optometric Center, Wyomissing, Pennsylvania
  - Optometry Group, PLLC, Memphis, Tennessee
  - Clarke Eyecare Center, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No